CLINICAL TRIAL: NCT06823713
Title: An Open-label Phase 1/2 Multicentre Study to Evaluate the Safety, Tolerability and Efficacy of RTX001 Autologous Macrophages in Participants With Liver Cirrhosis Who Have Hepatic Decompensation (EMERALD)
Brief Title: RTX001 Autologous Engineered Macrophages for Liver Cirrhosis
Acronym: EMERALD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Resolution Therapeutics Limited (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTX001-002; 2024-516288-10 (EudraCT Number)
Record Dates: First submitted 2024-11-06; First posted 2025-02-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: End-stage Liver Disease (ESLD); Cirrhosis, Liver; Cirrhosis, Decompensated; Liver Diseases; Fibrosis and Cirrhosis of Liver; Decompensated Liver Cirrhosis; Decompensated Cirrhosis; Steatotic Liver Disease
Keywords: Liver cirrhosis; Cirrhotic; Hepatic Cirrhosis; Chronic Liver Disease; Liver Fibrosis; Decompensated Liver Cirrhosis; Child-Pugh Score; MELD Score; Liver Function Tests; Hepatic Encephalopathy; End Stage Liver Disease (ESLD); Variceal Bleeding; Jaundice; Retractable Ascites; Autologous; Cell Therapy; Macrophage; Steatotic Liver Disease
MeSH Terms: conditions — End Stage Liver Disease; Liver Cirrhosis; Fibrosis; Liver Diseases; Hepatic Encephalopathy; Jaundice

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RTX001 (Experimental): Following the manufacture of RTX001, participants will be assigned into one of two groups based on the compensation status of their cirrhosis at this time as follows:
  * Stabilised Group: Participants who remain clinically stable, as assessed by the Investigator, since their qualifying decompensation event.
  * Subsequent Decompensation Group: Participants who have had a further decompensation event following their leukapheresis and/or the RTX001 manufacturing process.
  Treatment will be identical for both groups, and each participant will receive a maximum of four doses of RTX001 by intravenous infusion Patients in the Subsequent Decompensation Group need to have stabilised before receiving treatment.
  Interventions: Drug: RTX001

INTERVENTIONS:
Drug: RTX001 — RTX001 is an autologous engineered regenerative macrophage cell therapy

SUMMARY:
The purpose of this study is to assess the safety and efficacy of RTX001 in patients with end-stage liver disease. This study is the first time RTX001, a macrophage cell therapy engineered to have an anti-inflammatory and anti-fibrotic effect, will be given to humans.

DETAILED DESCRIPTION:
EMERALD is a first-in-human Phase 1/2 open label study designed to evaluate the safety, tolerability and efficacy of RTX001 in patients with end-stage liver disease following recent hepatic decompensation.

RTX001 is an autologous engineered macrophage cell therapy. It is made from a person's own cells. It uses a type of white blood cell called macrophages. These cells have been found to help improve liver function in participants with liver cirrhosis.

To produce RTX001, each study participant must first undergo steps that will allow us to collect white blood cells using a process called leukapheresis. Leukapheresis is a procedure in which white blood cells are separated from the collected blood using a specific machine. The collected white blood cells are sent to a manufacturing facility to make RTX001. As RTX001 is an autologous product, this means that it can only be given back to the same participant who donated the cells. The term "autologous macrophage" used in the study title refers to white blood cells (macrophages) coming from the same person's body (autologous).

The data in this study will be compared to the external control data from a Natural History Study called OPAL (NCT06380335) which is being conducted in a similar participant population from primarily the same study sites in the United Kingdom (UK) and EU.

ELIGIBILITY:
Individuals eligible to participate in this study must meet the following criteria:

Inclusion Criteria:

1. Male or female age ≥18-75 years.
2. Patient confirms willingness/ability to comply with all study procedures.
3. Diagnosis of liver cirrhosis based on at least one of:

   1. Clinical and radiological features that correlate with a diagnosis of cirrhosis.
   2. Transient elastography (Fibroscan) >15 kPa.
   3. Previous liver biopsy confirming histological features of cirrhosis.
4. Aetiology of liver disease of steatotic liver disease including MASLD or Met-ALD or ALD

   a. Participants with alcohol-related liver disease (ALD or Met-ALD) only if they are confirmed to not be drinking alcohol above Met-ALD limits defined in this protocol. (N.B. No more than 34% of the total treated participants in this protocol will be ALD [excludes Met-ALD]).
5. Hospitalised as an inpatient for a recent major hepatic decompensation event including ascites, hepatic encephalopathy, variceal bleed, HRS-AKI or SBP, this being the only hospitalisation for an hepatic decompensation event hospitalisation within the last 6 months, and where recent is defined as within 6 weeks of hospital discharge.
6. Outpatient: Medically refractory ascites (ONLY), that recurs (i.e., second therapeutic LVP) within a 6-month period. Medically refractory ascites is defined by the repeated (≥2) need for LVP (i.e., therapeutic, not diagnostic) at least once per 8 weeks despite best medical attempts to control the ascites by sodium restriction and diuretic treatment, as confirmed by the Investigator. Onset is defined as the date of the second therapeutic LVP.
7. Confirmatory PEth alcohol test <200 ng/ml
8. MELD score of 12-20 taken within two weeks of 'qualifying' decompensation event.
9. No known contradictions to filgrastim or leukapheresis procedure.
10. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
11. Willing and able to give signed informed consent, and if applicable assent.

Participants are excluded from the study if any of the following criteria apply:

Exclusion Criteria:

1. Liver cirrhosis due to:

   1. any viral hepatitidies, or
   2. autoimmune and cholestatic aetiologies including, but not limited to, primary biliary cholangitis and primary sclerosing cholangitis.
2. Acute liver disease in the absence of underlying liver cirrhosis, including, but not limited to, drug induced liver injury.
3. Any current organ failure requiring more than outpatient supportive care, and not associated with the participant's qualifying hepatic decompensation event.
4. Known splenomegaly ≥16 cm.
5. Thrombocytopenia <50×109/L.
6. Presence or suspicion of any of the following co-morbidities:

   1. History of liver transplantation or other organ transplant.
   2. ACLF.
   3. Sepsis (with positive microbial cultures) or as defined by the Principal Investigator, unless stable and is at least 4 weeks after having completed a full course of IV antibiotics.
   4. Known human immunodeficiency virus.
   5. Known syphilis.
   6. Known human T-lymphotropic virus 1.
   7. Pulmonary embolism.
   8. Hepatocellular carcinoma, or any active malignant disease within the last five years, (excluding non-melanoma skin cancer, cervical carcinoma in situ, superficial bladder cancer, benign polyps etc.).
   9. Co-hepatic morbidities e.g., portal vein thrombosis.
   10. Participants with hepatic hydrothorax are excluded unless it is a small hydrothorax, not clinically apparent, that is detected incidentally by radiologic evaluation that does not require clinical intervention.
   11. Chronic renal impairment (on dialysis) or unresolved AKI.
   12. Acute or chronic heart failure (New York Heart Association Grade III/IV).
   13. Porto-pulmonary hypertension.
   14. Severe chronic lung disease e.g., chronic obstructive pulmonary disease or interstitial lung disease where the forced expiratory volume in the first second (FEV1) is less than 50% and/or FEV1/forced vital capacity is less than 60%.
   15. Hepatopulmonary syndrome.
   16. Previous or current treatment with multiple infusions of albumin for therapeutic intent. [Use of albumin infusion at the time of large volume paracentesis for circulatory support is allowed.]
   17. Significant untreated/unstable psychiatric disease.
   18. Transjugular intrahepatic portosystemic shunt (TIPSS).
7. As judged by the Investigator, any evidence of intercurrent illness that is either life threatening or of clinical significance such that it might limit compliance with study procedures.
8. Current or planned use of immunomodulators or immunosuppressive medication; note: low doses of corticosteroids up to 10 mg/kg/day prednisone or equivalent are permitted, or inhaled steroids to manage asthma.
9. Received a gene or cell therapy at any time.
10. Current or planned use of a live attenuated vaccines four weeks or fewer prior to enrolment (and for 3 months after the last administered dose of RTX001).
11. Received any investigational product within the past 6 months, or five half-lives (whichever is longer) or participated in another investigational interventional study within 30 days prior to the screening visit.
12. Participants with a known hypersensitivity to dimethyl sulfoxide (DMSO).
13. Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
14. For female participants only - pregnant or breast-feeding or plans to become pregnant over the next year, or of childbearing potential and unwilling to comply with contraceptive requirements.
15. Alcohol misuse in the period between identification of the participant as potentially suitable for this study to Screening (Visit 1), defined as alcohol intake greater than three units/day for females and four units/day for males, or binge drinking (>14 units/day) as determined by the Investigator. N.B. One unit is equivalent to 14 g of alcohol: a half-pint (~240 mL) of beer, one glass (125 mL) of wine or one (25 mL) measure of spirits.
16. Intake of non-medically supervised drugs of abuse that are judged (by the Investigator) to be a high risk to the participants acute health or which makes the participant likely to be non-compliant with follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2028-08-29 (Estimated); Study Completion 2028-11-29 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | 2.5 years
  Incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs)
Safety and Tolerability | At each infusion; day of infusion up to two weeks post-infusion
  Incidence and severity of infusion reactions

SECONDARY OUTCOMES:
Time to clinical event | 2.5 years
  Time to clinical event, defined as all hepatic decompensation events including SBP and/or HRS-AKI, new listing for liver transplantation, liver transplantation, or death.
Time to mortality | 2.5 years
  Time-to all-cause mortality (hepatic related and all-cause).
Change in Model for End Stage Liver Disease score 3.0 (MELD3.0) | 2.5 years
  To evaluate changes in Model for End Stage Liver Disease (MELD3.0) scores, from baseline to end of study in the Stabilised Group participants.

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (8):
  - Bristol Royal Infirmary, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Royal Liverpool University Hospital, Liverpool
  - King's College Hospital, London
  - St George's Hospital, London
  - St Mary's Hospital, London
  - Nottingham University Hospital, Nottingham

REFERENCES:
- [Background] Forbes S et al., Hepatology. AASLD Abstract #0095 (2024)
- [Background] Brennan et al., Hepatology. AASLD Abstract #160 (2023) https://www.aasld.org/the-liver-meeting/open-label-parallel-group-phase-ii-randomised-controlled-trial-autologous
- [Background] LBP-007 Beneficial effects of autologous macrophage therapy on clinical outcomes in patients with compensated cirrhosis: extended follow-up data from a randomized controlled phase 2 trial Brennan, Paul et al. Journal of Hepatology, Volume 80, S81 DOI: 10.1016/S0168-8278(24)00574-9
- [Background] Moroni F, Dwyer BJ, Graham C, Pass C, Bailey L, Ritchie L, Mitchell D, Glover A, Laurie A, Doig S, Hargreaves E, Fraser AR, Turner ML, Campbell JDM, McGowan NWA, Barry J, Moore JK, Hayes PC, Leeming DJ, Nielsen MJ, Musa K, Fallowfield JA, Forbes SJ. Safety profile of autologous macrophage therapy for liver cirrhosis. Nat Med. 2019 Oct;25(10):1560-1565. doi: 10.1038/s41591-019-0599-8. Epub 2019 Oct 7. PMID 31591593
- See also: The OPAL Study on ClinicalTrials.gov — https://clinicaltrials.gov/study/NCT06380335
- See also: British Liver Trust - The EMERALD Study — https://britishlivertrust.org.uk/the-emerald-study/